CLINICAL TRIAL: NCT02304432
Title: Targeting a Genetic Mutation in Glycine Metabolism With D-cycloserine
Acronym: DCS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Principal Investigator, Deborah L. Levy, Director, Psychology Research Laboratory, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R21MH105732 (NIH)
Record Dates: First submitted 2014-11-26; First posted 2014-12-02 (Estimated); Results first posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: D-cycloserine; Glycine; Psychosis; Mutation; GABA
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Psychotic Disorders | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open label DCS (Experimental): Both participants received open label D-cycloserine (seromycin), 50 mg/d capsule for 8 weeks.
  Interventions: Drug: D-cycloserine
- DCS or placebo (Experimental): Randomized to DCS or placebo. Participants underwent double-blind placebo-controlled exposures to DCS for 6 weeks or placebo for 6 weeks. One participant received exposure to DCS for 6 weeks and then received placebo dosing for 6 weeks. The other participant received exposure to placebo dosing for 6 weeks and then DCS for 6 weeks.
  Interventions: Drug: D-cycloserine; Drug: DCS or placebo
- Second open label DCS (Experimental): Both participants received second open label exposures to D-cycloserine (seromycin), 50 mg/d capsule for 24 weeks.
  Interventions: Drug: D-cycloserine

INTERVENTIONS:
Drug: D-cycloserine — Both participants received open label D-cycloserine (seromycin), 50 mg/d capsule, x 8 weeks.
  Other Names: Seromycin (d-cycloserine)
  Arms: DCS or placebo; Open label DCS
Drug: DCS or placebo — Double-blind placebo-controlled exposures to DCS or placebo x 6 weeks. One participant received exposure to DCS x 6 weeks and then received placebo dosing x 6 weeks. The other participant received exposure to placebo dosing x 6 weeks and then DCS x 6 weeks.
  Other Names: Seromycin (d-cycloserine) or placebo
  Arms: DCS or placebo
Drug: D-cycloserine — Both participants received second open label D-cycloserine (seromycin), 50 mg/d capsule, x 8 weeks.
  Other Names: Seromycin (d-cycloserine)
  Arms: Second open label DCS

SUMMARY:
The purpose of this study is to assess the efficacy of d-cycloserine (DCS) as an augmentation strategy in two psychotic patients with a triplication (4 copies) of the glycine decarboxylase (GLDC) gene. Subjects will first undergo an eight-week open-label arm of treatment with DCS (50 mg/d) followed by six 6-week double-blind placebo-controlled exposures to DCS or placebo. The length of each double-blind arm is limited to six weeks to minimize the length of symptom exacerbation experienced by the subjects when they are receiving placebo. The randomization scheme will allow two consecutive exposures to DCS, but will not allow two consecutive exposures to placebo, again to minimize the length of any symptom exacerbation. At the end of the open-label DCS trial, the following procedures will be carried out: structural MRI (3T), proton 1H MRS (4T), fMRI (3T), steady-state auditory evoked potentials, and electroretinogram recordings. In addition, 1H MRS (4T) for 2 hours after a single oral dose of a DCS will be assessed. Baseline data on all of these measures were previously obtained as part of a different study registered in clinical trials.gov - NCT01720316). Positive, negative, and affective symptoms and neurocognitive function as well as plasma levels of large neutral and large and small neutral and excitatory amino acids and psychotropic drug levels will be assessed periodically. Pharmaceutical grade DCS) or placebo will be compounded and dispensed by the McLean Hospital Pharmacy.

The investigators hypothesize that mutation carriers will have reduced endogenous brain glycine and GABA levels and increased brain glutamate and glutamine levels. DCS administration will increase brain glycine in the two carriers compared to baseline and treatment with glycine (0.8g/kg).

The investigators hypothesize reduced activation of magnocellular pathways and abnormal ERPs modulated by NMDA in mutation carriers compared with non-carrier family members and controls.

. The investigators hypothesize that DCS, but not placebo, will improve positive, negative and affective symptoms as well as neurocognitive function.

The investigators also hypothesize that DCS will improve clinical and cognitive functioning, will partially normalize decreased baseline glycine and GABA and increased glutamate and glutamine, and will partially normalize magnocellular pathway activation and abnormal evoked potentials.

DETAILED DESCRIPTION:
Multiple rare structural variants of relatively recent evolutionary origin are recognized as important risk factors for schizophrenia (SZ) and other neurodevelopmental disorders (e.g., autism spectrum disorders, mental retardation, epilepsy) with odds ratios as high as 7-30. We have found a de novo structural rearrangement on chromosome 9p24.1 in two psychotic patients. One of the genes in this region is the gene encoding glycine decarboxylase (GLDC), which affects brain glycine metabolism. GLDC encodes the glycine decarboxylase or glycine cleavage system P-protein, which is involved in degradation of glycine in glia cells. Carriers of the GLDC triplication would be expected to have low levels of brain Gly, resulting in NMDA receptor-mediated hypofunction, which has been strongly implicated in the pathophysiology of schizophrenia.

There is an extensive literature on the effects of NMDA enhancing agents on positive, negative, and depressive symptoms and on neurocognitive function. Although many studies have reported positive results in at least one symptom domain, the results of other studies have been negative or ambiguous. Factors likely to contribute to this variability include: mechanism of action of the agent, compliance, concurrent treatment with first- vs second generation antipsychotic drugs, baseline glycine blood levels, presence/absence of kynurenine pathway metabolic abnormalities and individual differences in brain glycine uptake and metabolism . Genetic variants that impact the synthesis and breakdown of glycine, glutamate, or other modulators of NMDA receptor function are also likely to have significant effects. Although DCS augmentation has shown variable efficacy in patients unselected for having a mutation that would be expected to lower brain glycine levels, the GLDC triplication in the two carriers in this study would be expected to result in unusually low brain glycine levels, supporting its therapeutic potential as an augmentation strategy.

Thus, it is important to evaluate the therapeutic efficacy of DCS augmentation in individuals in whom there is a high prior probability of therapeutic benefit and to characterize the neurobiology of this mutation in terms of brain metabolites, brain function, and the pharmacokinetics of glycine metabolism using well-established methods.

ELIGIBILITY:
Inclusion Criteria:

* Carriers of a triplication in the glycine decarboxylase gene

Exclusion Criteria:

* Not carriers of a triplication in the glycine decarboxylase gene

Ages: 34 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09-27 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L. Levy, Ph.D., Principal Investigator — Mclean Hospital

REFERENCES:
- [Background] Sebat J, Levy DL, McCarthy SE. Rare structural variants in schizophrenia: one disorder, multiple mutations; one mutation, multiple disorders. Trends Genet. 2009 Dec;25(12):528-35. doi: 10.1016/j.tig.2009.10.004. Epub 2009 Oct 31. PMID 19883952
- [Background] Malhotra D, McCarthy S, Michaelson JJ, Vacic V, Burdick KE, Yoon S, Cichon S, Corvin A, Gary S, Gershon ES, Gill M, Karayiorgou M, Kelsoe JR, Krastoshevsky O, Krause V, Leibenluft E, Levy DL, Makarov V, Bhandari A, Malhotra AK, McMahon FJ, Nothen MM, Potash JB, Rietschel M, Schulze TG, Sebat J. High frequencies of de novo CNVs in bipolar disorder and schizophrenia. Neuron. 2011 Dec 22;72(6):951-63. doi: 10.1016/j.neuron.2011.11.007. PMID 22196331
- [Background] Heinzen EL, Radtke RA, Urban TJ, Cavalleri GL, Depondt C, Need AC, Walley NM, Nicoletti P, Ge D, Catarino CB, Duncan JS, Kasperaviciutey D, Tate SK, Caboclo LO, Sander JW, Clayton L, Linney KN, Shianna KV, Gumbs CE, Smith J, Cronin KD, Maia JM, Doherty CP, Pandolfo M, Duncan JS, Sander JW, Delanty N, Leppert D, Middleton LT, Gibson RA, Johnson MR, Matthews PM, Hosford D, Kalviainen R, Eriksson K, Kantanen A-M, Dorn T, Hansen J, Kramer G, Steinhoff BJ, Wieser H-G, Steinhoff BJ, Kramer G, Hansen J, Dorn T, Zumsteg D, Ortega M, Wood NW, Huxley-Jones J, Mikati M, Gallentine WB, Husain AM, Buckley PG, Stallings RL, Podgoreanu MV, Delanty N, Sisodiya SM, Goldstein DB. Rare deletions at 16p13.11 predispose to a diverse spectrum of sporadic epilepsy syndromes. Am J Hum Genet 2010;86:707-718.
- [Background] Weiss LA, Shen Y, Korn JM, Arking DE, Miller DT, Fossdal R, Saemundsen E, Stefansson H, Ferreira MA, Green T, Platt OS, Ruderfer DM, Walsh CA, Altshuler D, Chakravarti A, Tanzi RE, Stefansson K, Santangelo SL, Gusella JF, Sklar P, Wu BL, Daly MJ; Autism Consortium. Association between microdeletion and microduplication at 16p11.2 and autism. N Engl J Med. 2008 Feb 14;358(7):667-75. doi: 10.1056/NEJMoa075974. Epub 2008 Jan 9. PMID 18184952
- [Background] McCarthy S, Makarov V, Kirov G, Addington A, McClellan J, Yoon S, Perkins D, Dickel DE, Kusenda M, Krastoshevsky O, Krause V, Kumar RA, Grozeva D, Malhotra D, Walsh T, Zackai EH, Kaplan P, Ganesh J, Krantz ID, Spinner NB, Roccanova P, Bhandari A, Pavon K, Lakshmi B, Leotta A, Kendall J, Lee Y, Vacic V, Gary S, Iakoucheva L, Crow TJ, Christian SL, Lieberman J, Stroup S, Lehtimaki T, Puura K, Haldeman-Englert C, Pearl J, Goodell M, Willour VL, DeRosse P, Steele J, Kassem L, Wolff J, Chitkara N, McMahon F, Malhotra AK, Potash JB, Schulze T, Nothen MM, Cichon S, Rietschel M, Leibenluft E, Sutcliffe JS, Skuse D, Gill M, Gallagher L, Mendell NR, Consortium WTCC, Craddock N, Owen MJ, O'Donovan MC, Shaikh TH, Susser E, DeLisi LE, Sullivan PF, Deutsch CK, Rapoport J, Levy DL, King M-C, Sebat J. Microduplications of 16p11.2 are associated with schizophrenia. Nat Genet 2009;41:1223-1227.
- [Background] Olney JW, Farber NB. Glutamate receptor dysfunction and schizophrenia. Arch Gen Psychiatry. 1995 Dec;52(12):998-1007. doi: 10.1001/archpsyc.1995.03950240016004. PMID 7492260
- [Background] Coyle JT. Glutamate and schizophrenia: beyond the dopamine hypothesis. Cell Mol Neurobiol. 2006 Jul-Aug;26(4-6):365-84. doi: 10.1007/s10571-006-9062-8. Epub 2006 Jun 14. PMID 16773445
- [Background] Javitt DC. Glutamate and schizophrenia: phencyclidine, N-methyl-D-aspartate receptors, and dopamine-glutamate interactions. Int Rev Neurobiol. 2007;78:69-108. doi: 10.1016/S0074-7742(06)78003-5. PMID 17349858
- [Background] Tsai GE, Lin PY. Strategies to enhance N-methyl-D-aspartate receptor-mediated neurotransmission in schizophrenia, a critical review and meta-analysis. Curr Pharm Des. 2010;16(5):522-37. doi: 10.2174/138161210790361452. PMID 19909229
- [Background] Lin CH, Lane HY, Tsai GE. Glutamate signaling in the pathophysiology and therapy of schizophrenia. Pharmacol Biochem Behav. 2012 Feb;100(4):665-77. doi: 10.1016/j.pbb.2011.03.023. Epub 2011 Apr 1. PMID 21463651
- [Background] Heresco-Levy U, Javitt DC, Ermilov M, Mordel C, Horowitz A, Kelly D. Double-blind, placebo-controlled, crossover trial of glycine adjuvant therapy for treatment-resistant schizophrenia. Br J Psychiatry. 1996 Nov;169(5):610-7. doi: 10.1192/bjp.169.5.610. PMID 8932891
- [Background] Heresco-Levy U, Javitt DC, Ermilov M, Mordel C, Silipo G, Lichtenstein M. Efficacy of high-dose glycine in the treatment of enduring negative symptoms of schizophrenia. Arch Gen Psychiatry. 1999 Jan;56(1):29-36. doi: 10.1001/archpsyc.56.1.29. PMID 9892253
- [Background] Heresco-Levy U, Javitt DC. Comparative effects of glycine and D-cycloserine on persistent negative symptoms in schizophrenia: a retrospective analysis. Schizophr Res. 2004 Feb 1;66(2-3):89-96. doi: 10.1016/S0920-9964(03)00129-4. PMID 15061240
- [Background] Tsai G, Yang P, Chung LC, Lange N, Coyle JT. D-serine added to antipsychotics for the treatment of schizophrenia. Biol Psychiatry. 1998 Dec 1;44(11):1081-9. doi: 10.1016/s0006-3223(98)00279-0. PMID 9836012
- [Background] Tsai GE, Yang P, Chung LC, Tsai IC, Tsai CW, Coyle JT. D-serine added to clozapine for the treatment of schizophrenia. Am J Psychiatry. 1999 Nov;156(11):1822-5. doi: 10.1176/ajp.156.11.1822. PMID 10553752
- [Background] Tsai G, Lane HY, Yang P, Chong MY, Lange N. Glycine transporter I inhibitor, N-methylglycine (sarcosine), added to antipsychotics for the treatment of schizophrenia. Biol Psychiatry. 2004 Mar 1;55(5):452-6. doi: 10.1016/j.biopsych.2003.09.012. PMID 15023571
- [Background] Tsai GE, Yang P, Chang YC, Chong MY. D-alanine added to antipsychotics for the treatment of schizophrenia. Biol Psychiatry. 2006 Feb 1;59(3):230-4. doi: 10.1016/j.biopsych.2005.06.032. Epub 2005 Sep 9. PMID 16154544
- [Background] Javitt DC, Silipo G, Cienfuegos A, Shelley AM, Bark N, Park M, Lindenmayer JP, Suckow R, Zukin SR. Adjunctive high-dose glycine in the treatment of schizophrenia. Int J Neuropsychopharmacol. 2001 Dec;4(4):385-91. doi: 10.1017/S1461145701002590. PMID 11806864
- [Background] Goff DC, Tsai G, Manoach DS, Flood J, Darby DG, Coyle JT. D-cycloserine added to clozapine for patients with schizophrenia. Am J Psychiatry. 1996 Dec;153(12):1628-30. doi: 10.1176/ajp.153.12.1628. PMID 8942463
- [Background] Lane HY, Liu YC, Huang CL, Chang YC, Liau CH, Perng CH, Tsai GE. Sarcosine (N-methylglycine) treatment for acute schizophrenia: a randomized, double-blind study. Biol Psychiatry. 2008 Jan 1;63(1):9-12. doi: 10.1016/j.biopsych.2007.04.038. Epub 2007 Jul 20. PMID 17659263
- [Background] Goff DC, Henderson DC, Evins AE, Amico E. A placebo-controlled crossover trial of D-cycloserine added to clozapine in patients with schizophrenia. Biol Psychiatry. 1999 Feb 15;45(4):512-4. doi: 10.1016/s0006-3223(98)00367-9. PMID 10071726
- [Background] Evins AE, Fitzgerald SM, Wine L, Rosselli R, Goff DC. Placebo-controlled trial of glycine added to clozapine in schizophrenia. Am J Psychiatry. 2000 May;157(5):826-8. doi: 10.1176/appi.ajp.157.5.826. PMID 10784481
- [Background] van Berckel BN, Evenblij CN, van Loon BJ, Maas MF, van der Geld MA, Wynne HJ, van Ree JM, Kahn RS. D-cycloserine increases positive symptoms in chronic schizophrenic patients when administered in addition to antipsychotics: a double-blind, parallel, placebo-controlled study. Neuropsychopharmacology. 1999 Aug;21(2):203-10. doi: 10.1016/S0893-133X(99)00014-7. PMID 10432468
- [Background] Wonodi I, Schwarcz R. Cortical kynurenine pathway metabolism: a novel target for cognitive enhancement in Schizophrenia. Schizophr Bull. 2010 Mar;36(2):211-8. doi: 10.1093/schbul/sbq002. Epub 2010 Feb 10. PMID 20147364
- [Background] Erhardt S, Schwieler L, Nilsson L, Linderholm K, Engberg G. The kynurenic acid hypothesis of schizophrenia. Physiol Behav. 2007 Sep 10;92(1-2):203-9. doi: 10.1016/j.physbeh.2007.05.025. Epub 2007 May 21. PMID 17573079
- [Background] Kaufman MJ, Prescot AP, Ongur D, Evins AE, Barros TL, Medeiros CL, Covell J, Wang L, Fava M, Renshaw PF. Oral glycine administration increases brain glycine/creatine ratios in men: a proton magnetic resonance spectroscopy study. Psychiatry Res. 2009 Aug 30;173(2):143-9. doi: 10.1016/j.pscychresns.2009.03.004. Epub 2009 Jun 24. PMID 19556112
- [Background] Buchanan RW, Javitt DC, Marder SR, Schooler NR, Gold JM, McMahon RP, Heresco-Levy U, Carpenter WT. The Cognitive and Negative Symptoms in Schizophrenia Trial (CONSIST): the efficacy of glutamatergic agents for negative symptoms and cognitive impairments. Am J Psychiatry. 2007 Oct;164(10):1593-602. doi: 10.1176/appi.ajp.2007.06081358. PMID 17898352
- [Background] Goff DC, Tsai G, Levitt J, Amico E, Manoach D, Schoenfeld DA, Hayden DL, McCarley R, Coyle JT. A placebo-controlled trial of D-cycloserine added to conventional neuroleptics in patients with schizophrenia. Arch Gen Psychiatry. 1999 Jan;56(1):21-7. doi: 10.1001/archpsyc.56.1.21. PMID 9892252
- [Background] Goff DC, Herz L, Posever T, Shih V, Tsai G, Henderson DC, Freudenreich O, Evins AE, Yovel I, Zhang H, Schoenfeld D. A six-month, placebo-controlled trial of D-cycloserine co-administered with conventional antipsychotics in schizophrenia patients. Psychopharmacology (Berl). 2005 Apr;179(1):144-50. doi: 10.1007/s00213-004-2032-2. Epub 2004 Oct 21. PMID 15502972
- [Background] Goff DC, Cather C, Gottlieb JD, Evins AE, Walsh J, Raeke L, Otto MW, Schoenfeld D, Green MF. Once-weekly D-cycloserine effects on negative symptoms and cognition in schizophrenia: an exploratory study. Schizophr Res. 2008 Dec;106(2-3):320-7. doi: 10.1016/j.schres.2008.08.012. Epub 2008 Sep 16. PMID 18799288
- [Background] Heresco-Levy U, Javitt DC, Ermilov M, Silipo G, Shimoni J. Double-blind, placebo-controlled, crossover trial of D-cycloserine adjuvant therapy for treatment-resistant schizophrenia. Int J Neuropsychopharmacol. 1998 Dec;1(2):131-135. doi: 10.1017/S1461145798001242. PMID 11281957
- [Background] Heresco-Levy U, Ermilov M, Shimoni J, Shapira B, Silipo G, Javitt DC. Placebo-controlled trial of D-cycloserine added to conventional neuroleptics, olanzapine, or risperidone in schizophrenia. Am J Psychiatry. 2002 Mar;159(3):480-2. doi: 10.1176/appi.ajp.159.3.480. PMID 11870017
- [Background] Prescot AP, de B Frederick B, Wang L, Brown J, Jensen JE, Kaufman MJ, Renshaw PF. In vivo detection of brain glycine with echo-time-averaged (1)H magnetic resonance spectroscopy at 4.0 T. Magn Reson Med. 2006 Mar;55(3):681-6. doi: 10.1002/mrm.20807. PMID 16453318
- [Background] Martinez A, Hillyard SA, Dias EC, Hagler DJ Jr, Butler PD, Guilfoyle DN, Jalbrzikowski M, Silipo G, Javitt DC. Magnocellular pathway impairment in schizophrenia: evidence from functional magnetic resonance imaging. J Neurosci. 2008 Jul 23;28(30):7492-500. doi: 10.1523/JNEUROSCI.1852-08.2008. PMID 18650327
- [Background] Butler PD, Schechter I, Zemon V, Schwartz SG, Greenstein VC, Gordon J, Schroeder CE, Javitt DC. Dysfunction of early-stage visual processing in schizophrenia. Am J Psychiatry. 2001 Jul;158(7):1126-33. doi: 10.1176/appi.ajp.158.7.1126. PMID 11431235
- [Background] Jensen JE, Licata SC, Ongur D, Friedman SD, Prescot AP, Henry ME, Renshaw PF. Quantification of J-resolved proton spectra in two-dimensions with LCModel using GAMMA-simulated basis sets at 4 Tesla. NMR Biomed. 2009 Aug;22(7):762-9. doi: 10.1002/nbm.1390. PMID 19388001
- [Background] Ongur D, Jensen JE, Prescot AP, Stork C, Lundy M, Cohen BM, Renshaw PF. Abnormal glutamatergic neurotransmission and neuronal-glial interactions in acute mania. Biol Psychiatry. 2008 Oct 15;64(8):718-726. doi: 10.1016/j.biopsych.2008.05.014. Epub 2008 Jul 7. PMID 18602089
- [Result] Duncan EJ, Szilagyi S, Schwartz MP, Bugarski-Kirola D, Kunzova A, Negi S, Stephanides M, Efferen TR, Angrist B, Peselow E, Corwin J, Gonzenbach S, Rotrosen JP. Effects of D-cycloserine on negative symptoms in schizophrenia. Schizophr Res. 2004 Dec 1;71(2-3):239-48. doi: 10.1016/j.schres.2004.03.013. PMID 15474895
- [Derived] Bodkin JA, Coleman MJ, Godfrey LJ, Carvalho CMB, Morgan CJ, Suckow RF, Anderson T, Ongur D, Kaufman MJ, Lewandowski KE, Siegel AJ, Waldstreicher E, Grochowski CM, Javitt DC, Rujescu D, Hebbring S, Weinshilboum R, Rodriguez SB, Kirchhoff C, Visscher T, Vuckovic A, Fialkowski A, McCarthy S, Malhotra D, Sebat J, Goff DC, Hudson JI, Lupski JR, Coyle JT, Rudolph U, Levy DL. Targeted Treatment of Individuals With Psychosis Carrying a Copy Number Variant Containing a Genomic Triplication of the Glycine Decarboxylase Gene. Biol Psychiatry. 2019 Oct 1;86(7):523-535. doi: 10.1016/j.biopsych.2019.04.031. Epub 2019 May 9. PMID 31279534

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First, Then DCS: One of the sequences during the DB period; dose of DCS, freq of admin; length of trial
  Randomized to DCS or placebo. Participants underwent double-blind placebo-controlled exposures to DCS for 6 weeks or placebo for 6 weeks. One participant received exposure to DCS for 6 weeks and then received placebo dosing for 6 weeks. The other participant received exposure to placebo dosing for 6 weeks and then DCS for 6 weeks.
  D-cycloserine: Both participants received open label D-cycloserine (seromycin), 50 mg/d capsule, x 8 weeks.
  DCS or placebo: Double-blind placebo-controlled exposures to DCS or placebo x 6 weeks. One participant received exposure to DCS x 6 weeks and then received placebo dosing x 6 weeks. The other participant received exposure to placebo dosing x 6 weeks and then DCS x 6 weeks.
- DCS First, Then Placebo: One of the sequences during the DB period; dose of DCS, freq of admin; length of trial
Period: Open Label DCS
Arm/Group | Open Label DCS | Placebo First, Then DCS | DCS First, Then Placebo | Second Open Label DCS
Started | 2 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Double-Blind DCS Placebo Crossover
Arm/Group | Open Label DCS | Placebo First, Then DCS | DCS First, Then Placebo | Second Open Label DCS
Started | 0 | 1 | 1 | 0
Completed | 0 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Second Open Label DCS
Arm/Group | Open Label DCS | Placebo First, Then DCS | DCS First, Then Placebo | Second Open Label DCS
Started | 0 | 0 | 0 | 2
Completed | 0 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Both participants received open label D-cycloserine (seromycin), 50 mg/d capsule for 8 weeks.
  D-cycloserine: Both participants received open label D-cycloserine (seromycin), 50 mg/d capsule, x 8 weeks.
  Add crossover phase and second OL phase
Arm/Group | All Study Participants
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] — age at beginning of study
  years | 42 [34 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Symptom Scores
Description: Positive and Negative Symptom Scale (PANSS) measures positive and negative symptoms of schizophrenia. The sum of ratings for seven positive symptoms is measured on a scale from 7-49 with 7 meaning no symptoms and 49 meaning severe symptoms.The sum of ratings for seven negative symptoms is measured on a scale from 7-49 with 7 meaning no symptoms and 49 meaning severe symptoms.
Time Frame: Baseline & at 2, 4, 6 & 8 Weeks during open-label phase 1 and every 2 weeks up to 24 weeks during open label phase 2
Measure: Median (Full Range); unit: units on a scale
Groups:
- First Open Label DCS: Both participants received first open label exposure to D-cycloserine (seromycin), 50 mg/d capsule, for 8 weeks.
- Second Open Label DCS: Both participants received second open label exposure to D-cycloserine (seromycin), 50 mg/d capsule, for 24 weeks.
Arm/Group | First Open Label DCS | Second Open Label DCS
Number analyzed (Participants) | 2 | 2
units on a scale
  Baseline positive | 14.5 [12 to 17] | 11 [9 to 13]
  Baseline negative | 14.5 [11 to 18] | 14 [11 to 17]
  2 weeks positive | 10 [9 to 11] | 11 [9 to 13]
  2 weeks negative | 12 [9 to 15] | 14 [11 to 17]
  4 weeks positive | 10.5 [10 to 11] | 10.5 [9 to 12]
  4 weeks negative | 12 [9 to 15] | 13.5 [11 to 16]
  6 weeks positive | 9 [8 to 10] | 9 [8 to 10]
  6 weeks negative | 12 [9 to 15] | 13 [11 to 15]
  8 weeks positive | 9 [8 to 10] | 9.5 [8 to 11]
  8 weeks negative | 12 [9 to 15] | 12 [9 to 15]
  10 weeks positive | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 10.5 [10 to 11]
  10 weeks negative | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 13 [11 to 15]
  12 weeks positive | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 11 [9 to 13]
  12 weeks negative | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 12 [9 to 15]
  14 weeks positive | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 10 [8 to 12]
  14 weeks negative | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 12 [9 to 15]
  16 weeks positive | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 10.5 [10 to 11]
  16 weeks negative | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 12 [9 to 15]
  18 weeks positive | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 10.5 [9 to 12]
  18 weeks negative | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 12 [9 to 15]
  20 weeks positive | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 10.5 [9 to 12]
  20 weeks negative | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 12 [9 to 15]
  22 weeks positive | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 9.5 [8 to 11]
  22 weeks negative | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 12 [9 to 15]
  24 weeks positive | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 10 [8 to 12]
  24 weeks negative | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 12 [9 to 15]

2. Primary Outcome: Positive and Negative Symptom Scores
Description: as for outcome 1
Time Frame: Baseline, 2, 4, & 6 weeks (crossover periods)
Measure: Number; unit: units on a scale
Arm/Group | Placebo First, Then DCS | DCS First, Then Placebo
Number analyzed (Participants) | 1 | 1
units on a scale
  Baseline positive for first intervention | 11 | 10
  Baseline negative symptoms for first intervention | 9 | 15
  2 weeks positive for first intervention | 12 | 10
  2 weeks negative for first intervention | 15 | 15
  4 weeks positive for first intervention | 11 | 10
  4 weeks negative for first intervention | 13 | 15
  6 weeks positive for first intervention | 13 | 10
  6 weeks negative for first intervention | 13 | 15
  Baseline positive for second intervention | 13 | 15
  Baseline negative for second intervention | 13 | 18
  2 weeks positive for second intervention | 10 | 15
  2 weeks negative for second intervention | 11 | 18
  4 weeks positive for second intervention | 9 | 15
  4 weeks negative for second intervention | 11 | 18
  6 weeks positive for second intervention | 9 | 14
  6 weeks negative for second intervention | 11 | 18

3. Primary Outcome: Brief Psychiatric Rating Scale (BPRS) Scores
Description: Total BPRS score measures severity of 18 psychiatric symptoms. Each symptom is scored 1-7 with the total score ranging from 18-126. 18 means no symptoms and 126 means very severe symptoms.
Time Frame: Baseline & at 2, 4, 6 & 8 Weeks during open-label phase 1 and every 2 weeks up to 24 weeks during open label phase 2
Measure: Median (Full Range); unit: units on a scale
Groups:
- First Open Label DCS: Both participants received open label D-cycloserine (seromycin), 50 mg/d capsule, for 8 weeks.
Arm/Group | First Open Label DCS | Second Open Label DCS
Number analyzed (Participants) | 2 | 2
units on a scale
  Baseline BPRS | 37 [34 to 40] | 31.5 [28 to 35]
  2 weeks BPRS | 25 [22 to 28] | 30.5 [27 to 34]
  4 weeks BPRS | 26 [24 to 28] | 28 [27 to 29]
  6 weeks BPRS | 24 [22 to 26] | 25.5 [25 to 26]
  8 weeks BPRS | 24.5 [23 to 26] | 26 [24 to 28]
  10 weeks BPRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 26.5 [26 to 27]
  12 weeks BPRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 26 [24 to 28]
  14 weeks BPRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 25.5 [24 to 27]
  16 weeks BPRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 28.5 [27 to 30]
  18 weeks BPRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 27 [25 to 29]
  20 weeks BPRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 25 [23 to 27]
  22 weeks BPRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 24.5 [22 to 27]
  24 weeks BPRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 26.5 [25 to 28]

4. Primary Outcome: Brief Psychiatric Rating Scale (BPRS) Scores
Description: as for outcome 3
Time Frame: Baseline, 2, 4, & 6 weeks (crossover periods)
Measure: Number; unit: units on a scale
Arm/Group | Placebo First, Then DCS | DCS First, Then Placebo
Number analyzed (Participants) | 1 | 1
units on a scale
  Baseline BPRS for first intervention | 29 | 26
  2 weeks BPRS for first intervention | 35 | 25
  4 weeks BPRS for first intervention | 33 | 25
  6 weeks BPRS for first intervention | 35 | 26
  Baseline BPRS for second intervention | 36 | 39
  2 weeks BPRS for second intervention | 30 | 45
  4 weeks BPRS for second intervention | 27 | 45
  6 weeks BPRS for second intervention | 28 | 38

5. Primary Outcome: Clinical Global Impression (CGI) Severity Scores
Description: CGI severity scores measure severity of mental illness on a scale of 1-7 where 1 means normal, not at all ill, 2 means borderline mentally ill, 3 means mildly ill, 4 means moderately ill, 5 means markedly ill, 6 means severely ill and 7 means among the most extremely ill patients.
Time Frame: Baseline & at 2, 4, 6 & 8 Weeks during open-label phase 1 and every 2 weeks up to 24 weeks during open label phase 2
Measure: Median (Full Range); unit: units on a scale
Groups:
- Second Open Label DCS: Both participants received second open label exposures to D-cycloserine (seromycin), 50 mg/d capsule, for 24 weeks.
Arm/Group | First Open Label DCS | Second Open Label DCS
Number analyzed (Participants) | 2 | 2
units on a scale
  Baseline CGI | 4 [4 to 4] | 2.5 [2 to 3]
  2 weeks CGI | 2 [2 to 2] | 2.5 [2 to 3]
  4 weeks CGI | 2 [2 to 2] | 2.5 [2 to 3]
  6 weeks CGI | 2 [2 to 2] | 2.5 [2 to 3]
  8 weeks CGI | 2 [2 to 2] | 2.5 [2 to 3]
  10 weeks CGI | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 3 [3 to 3]
  12 weeks CGI | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 2.5 [2 to 3]
  14 weeks CGI | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 2 [2 to 2]
  16 weeks CGI | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 2.5 [2 to 3]
  18 weeks CGI | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 2.5 [2 to 3]
  20 weeks CGI | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 2.5 [2 to 3]
  22 weeks CGI | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 2.5 [2 to 3]
  24 weeks CGI | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 2.5 [2 to 3]

6. Primary Outcome: Clinical Global Impression (CGI) Severity Scores
Description: as for outcome 5
Time Frame: Baseline, 2, 4, & 6 weeks (crossover periods)
Measure: Number; unit: units on a scale
Arm/Group | Placebo First, Then DCS | DCS First, Then Placebo
Number analyzed (Participants) | 1 | 1
units on a scale
  Baseline CGI for first intervention | 1 | 2
  2 weeks CGI for first intervention | 3 | 2
  4 weeks CGI for first intervention | 3 | 2
  6 weeks CGI for first intervention | 3 | 2
  Baseline CGI for second intervention | 3 | 3
  2 weeks CGI for second intervention | 2 | 3
  4 weeks CGI for second intervention | 2 | 3
  6 weeks CGI for second intervention | 2 | 3

7. Primary Outcome: Mania Symptom Scores
Description: Young Mania Rating Scale (YMRS) measures severity of manic symptoms. The sum of the ratings for 7 symptoms of mania is measured on a scale of 0-4 and the sumof 4 symptoms of mania is measured on a scale of 0-8 to yield a total score ranging from 0-60, with 0 meaning no manic symptoms and 60 meaning severe manic symptoms.
Time Frame: Baseline & at 2, 4, 6 & 8 Weeks during open-label phase 1 and every 2 weeks up to 24 weeks during open label phase 2
Measure: Median (Full Range); unit: units on a scale
Arm/Group | First Open Label DCS | Second Open Label DCS
Number analyzed (Participants) | 2 | 2
units on a scale
  Baseline YMRS | 2 [2 to 2] | 0 [0 to 0]
  2 weeks YMRS | 1 [0 to 2] | 0 [0 to 0]
  4 weeks YMRS | 1 [0 to 2] | 0 [0 to 0]
  6 weeks YMRS | 0 [0 to 0] | 0 [0 to 0]
  8 weeks YMRS | 0 [0 to 0] | 0 [0 to 0]
  10 weeks YMRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 0 [0 to 0]
  12 weeks YMRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 0 [0 to 0]
  14 weeks YMRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 0 [0 to 0]
  16 weeks YMRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 0 [0 to 0]
  18 weeks YMRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 0 [0 to 0]
  20 weeks YMRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 0 [0 to 0]
  22 weeks YMRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 0 [0 to 0]
  24 weeks YMRS | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 1 [0 to 2]

8. Primary Outcome: Depression Symptom Scores
Description: Hamilton Depression Scale (HAM) measures severity of depression symptoms. The sum of the ratings for 9 depression symptoms is measured on a scale of 0-2 with 0 meaning no depression symptoms and 2 meaning some level of severity of that specific symptom. The rating for one depression symptom is measured on a scale of 0-3 with 0 meaning no depression symptoms and 3 meaning a severe level of that specific symptom. The sum of ratings for 11 depression symptoms is measured on a scale of 0-4, with 0 meaning no symptoms and 4 meaning a severe level of that specific symptom. The three sums are added to produce an overall depression rating scale score ranging from 0-65. Higher scores indicate worse depression symptoms.
Time Frame: Baseline & at 2, 4, 6 & 8 Weeks during open-label phase 1 and every 2 weeks up to 24 weeks during open label phase 2
Measure: Median (Full Range); unit: units on a scale
Arm/Group | First Open Label DCS | Second Open Label DCS
Number analyzed (Participants) | 2 | 2
units on a scale
  Baseline HAM | 5 [4 to 6] | 0.5 [0 to 1]
  2 weeks HAM | 1.5 [0 to 3] | 1 [1 to 1]
  4 weeks HAM | 1 [0 to 2] | 1 [0 to 2]
  6 weeks HAM | 0.5 [0 to 1] | 0 [0 to 0]
  8 weeks HAM | 1.5 [0 to 3] | 2.5 [0 to 5]
  10 weeks HAM | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 0 [0 to 0]
  12 weeks HAM | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 0 [0 to 0]
  14 weeks HAM | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 0 [0 to 0]
  16 weeks HAM | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 3.5 [0 to 7]
  18 weeks HAM | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 0 [0 to 0]
  20 weeks HAM | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 0 [0 to 0]
  22 weeks HAM | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 0 [0 to 0]
  24 weeks HAM | NA [NA to NA] — This open label period lasted only 8 weeks, so no additional data were collected for this time point. | 0 [0 to 0]

9. Primary Outcome: Mania Symptom Scores
Description: as for outcome 7
Time Frame: Baseline, 2, 4, & 6 weeks (crossover periods)
Measure: Number; unit: units on a scale
Arm/Group | Placebo First, Then DCS | DCS First, Then Placebo
Number analyzed (Participants) | 1 | 1
units on a scale
  Baseline YMRS for first intervention | 1 | 0
  2 weeks YMRS for first intervention | 0 | 0
  4 weeks YMRS for first intervention | 0 | 0
  6 weeks YMRS for first intervention | 0 | 0
  Baseline YMRS for second intervention | 4 | 0
  2 weeks YMRS for second intervention | 1 | 0
  4 weeks YMRS for second intervention | 1 | 0
  6 weeks YMRS for second intervention | 1 | 0

10. Primary Outcome: Depression Symptom Scores
Description: as for outcome 8
Time Frame: Baseline, 2, 4, & 6 weeks (crossover periods)
Measure: Number; unit: units on a scale
Arm/Group | Placebo First, Then DCS | DCS First, Then Placebo
Number analyzed (Participants) | 1 | 1
units on a scale
  Baseline HAM for first intervention | 4 | 0
  2 weeks HAM for first intervention | 5 | 1
  4 weeks HAM for first intervention | 2 | 0
  6 weeks HAM for first intervention | 10 | 0
  Baseline HAM for second intervention | 0 | 2
  2 weeks HAM for second intervention | 0 | 12
  4 weeks HAM for second intervention | 0 | 9
  6 weeks HAM for second intervention | 0 | 2

11. Secondary Outcome: Neurocognitive Function
Description: Scores on each of 8 domains of cognitive function (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning/problem solving, social cognition, overall composite). Scores are T scores ranging from 0-100, with 50 representing the mean for a population based on a normal distribution, standard deviation of 10. Higher scores signify better functioning.
Time Frame: Baseline and Week 8 of open-label DCS treatment
Population: The on DCS data were collected during week 8 of the first open-label portion of the study in one subject and in week 8 of the second open-label portion of the study in the other subject for logistical reasons.
Measure: Median (Full Range); unit: T scores
Groups:
- Open Label DCS: During the first open label period, both participants received D-cycloserine (seromycin), 50 mg/d capsule, for 8 weeks. During the second open-label period, both participants received D-cycloserine (seromycin), 50 mg/d capsule, for 24 weeks. One subject was tested at the beginning of week 8 of the first open-label period and the other subject was tested at the beginning of week 8 of the second open-label period.
Arm/Group | Open Label DCS
Number analyzed (Participants) | 2
T scores
  Baseline Processing Speed | 48.5 [43 to 54]
  Baseline Attention/Vigilance | 44.5 [39 to 50]
  Baseline Working Memory | 38.5 [38 to 39]
  Baseline Verbal Learning | 54 [45 to 63]
  Baseline Visual Learning | 50.5 [50 to 51]
  Baseline Reasoning/Problem Solving | 52.5 [52 to 53]
  Baseline Social Cognition | 48 [44 to 52]
  Baseline Overall Composite Score | 46.5 [45 to 48]
  Week 8 of open-label DCS Processing Speed | 52.5 [51 to 54]
  Week 8 of open-label DCS Attention/Vigilance | 47.5 [39 to 56]
  Week 8 of open-label DCS Working Memory | 50.5 [49 to 52]
  Week 8 of open-label DCS Verbal Learning | 43.5 [42 to 45]
  Week 8 of open-label DCS Visual Learning | 54.5 [51 to 58]
  Week 8 of open-label DCS Reasoning/Problem Solving | 66.5 [65 to 68]
  Week 8 of open-label DCS Social Cognition | 44.5 [42 to 47]
  Week 8 of open-label DCS Overall Composite Score | 51.5 [49 to 54]

12. Secondary Outcome: Brain Glycine/CR Ratio
Description: Proton magnetic resonance spectroscopy at 4T: brain glycine/CR ratio. Participants were assessed at baseline (pre-glycine challenge dose and 60, 80, 100 and 120 minutes post glycine dose) and in week 8 of of open-label DCS treatment: pre-DCS dose, and 60, 80, 100 and 120 minutes post DCS dose. Measured in posterior occipital cortex.
Time Frame: Baseline and Week 8 of DCS treatment
Population: Data collected only during only one of the open label periods for financial and logistical reasons. Data were collected in week 8 of the first open-label DCS exposure in one subject and in week 8 of the second open-label DCS exposure in the other subject for logistical reasons.
Measure: Median (Full Range); unit: ratio
Groups:
- Open Label DCS: During the first open label period, both participants received D-cycloserine (seromycin), 50 mg/d capsule, for 8 weeks. During the second open-label period, both participants received D-cycloserine (seromycin), 50 mg/d capsule, for 24 weeks. OOne subject was tested at the beginning of week 8 of the first open-label period and the other subject was tested at the beginning of week 8 of the second open-label period.
Arm/Group | Open Label DCS
Number analyzed (Participants) | 2
ratio
  Baseline | 0.41245 [0.2558 to 0.5691]
  Baseline at 60 minutes | 0.50375 [0.3918 to 0.6157]
  Baseline at 80 minutes | 0.65295 [0.6428 to 0.6631]
  Baseline at 100 minutes | 0.61505 [0.5938 to 0.6363]
  Baseline at 120 minutes | 0.8256 [0.6953 to 0.9559]
  Week 8 of DCS: Baseline | 0.10977 [0.00007 to 0.21947]
  Week 8 of DCS: 60 minutes | 0.248885 [0.24294 to 0.25483]
  Week 8 of DCS: 80 minutes | 0.32609 [0.24571 to 0.40647]
  Week 8 of DCS: 100 minutes | 0.32052 [0.24289 to 0.39815]
  Week 8 of DCS: 120 minutes | 0.312155 [0.1903 to 0.43401]

13. Secondary Outcome: Auditory Evoked Potentials in Latency (Msec)
Description: Auditory evoked potential latency: P300 at fz, cz, and pz; N100 at fz and cz; P200 at fz and cz.
Time Frame: Baseline and Week 8 of DCS treatment
Population: Only one subject had normal hearing, which is required for valid data collection.
Measure: Number; unit: msec
Groups:
- First Open Label DCS: The subject received the first open label exposure to D-cycloserine (seromycin), 50 mg/d capsule, for 8 weeks and was tested at the beginning of week 8.
Arm/Group | First Open Label DCS
Number analyzed (Participants) | 1
msec
  P300 at fz: Baseline | 279.297
  P300 at cz: Baseline | 279.297
  P300 at pz: Baseline | 279.297
  N100 at fz: Baseline | 97.656
  N100 at cz: Baseline | 91.797
  P200 at fz: Baseline | 197.266
  P200 at cz: Baseline | 193.359
  P300 at fz: Week 8 of DCS | 294.920
  P300 at cz: Week 8 of DCS | 294.000
  P300 at pz: Week 8 of DCS | 294
  N100 at fz: Week 8 of DCS | 87.9
  N100 at cz: Week 8 of DCS | 88.000
  P200 at fz: Week 8 of DCS | 212.890
  P200 at cz: Week 8 of DCS | 212.000

14. Secondary Outcome: Auditory Evoked Potentials in Amplitude (Degrees Measured in Microvolts)
Description: Auditory evoked potential amplitude: P300 at fz, cz, and pz; N100 at fz and cz; P200 at fz and cz; P50 S1 and S2; mismatch negativity (MMN) at fz and cz.
Time Frame: Baseline and Week 8 of DCS treatment
Population: Only one subject had normal hearing, which is required for valid data collection.
Measure: Number; unit: microvolts
Arm/Group | First Open Label DCS
Number analyzed (Participants) | 1
microvolts
  P300 at fz: Baseline | -0.635
  P300 at cz: Baseline | 6.529
  P300 at pz: Baseline | 5.340
  N100 at fz: Baseline | -3.926
  N100 at cz: Baseline | -3.615
  P200 at fz: Baseline | 1.662
  P200 at cz: Baseline | 6.591
  P50 S1: Baseline | 2.759
  P50 S2: Baseline | 1.23
  MMN at fz: Baseline | -3.356
  MMN at cz: Baseline | -4.130
  P300 at fz: Week 8 of DCS | 3.030
  P300 at cz: Week 8 of DCS | 6.810
  P300 at pz: Week 8 of DCS | 6.620
  N100 at fz: Week 8 of DCS | -3.260
  N100 at cz: Week 8 of DCS | -3.940
  P200 at fz: Week 8 of DCS | 8.200
  P200 at cz: Week 8 of DCS | 8.160
  P50 S1: Week 8 of DCS | 1.36
  P50 S2: Week 8 of DCS | 0.4
  MMN at fz: Week 8 of DCS | -3.330
  MMN at cz: Week 8 of DCS | -1.540

15. Secondary Outcome: Auditory Evoked Potentials in Gamma Oscillations (the Power Spectrum is Measured in Microvolts Squared)
Description: Auditory evoked potential gamma: G40 hz phase locking at fz and cz; G30 hz phase locking at fz and cz; G20 hz phase locking at fz and cz
Time Frame: Baseline and Week 8 of DCS treatment
Population: Only one subject had normal hearing, which is required for valid data collection.
Measure: Number; unit: microvolts squared
Arm/Group | First Open Label DCS
Number analyzed (Participants) | 1
microvolts squared
  G40 hz phase locking at fz: Baseline | 0.135
  G40 hz phase locking at cz: Baseline | 0.168
  G30 hz phase locking at fz: Baseline | 0.190
  G30 hz phase locking at cz: Baseline | 0.163
  G20 hz phase locking at fz: Baseline | 0.023
  G20 hz phase locking at cz: Baseline | 0.030
  G40 hz phase locking at fz: Week 8 of DCS | 0.344
  G40 hz phase locking at cz: Week 8 of DCS | 0.381
  G30 hz phase locking at fz: Week 8 of DCS | 0.168
  G30 hz phase locking at cz: Week 8 of DCS | 0.19
  G20 hz phase locking at fz: Week 8 of DCS | 0.01
  G20 hz phase locking at cz: Week 8 of DCS | -0.01

16. Secondary Outcome: Auditory Evoked Potentials - P50 Ratio (P50 S2/S1) (Amplitude)
Description: Auditory evoked potential amplitude: P50 ratio (P50 S2/S1)
Time Frame: Baseline and Week 8 of DCS treatment
Population: Only one subject had normal hearing, which is required for valid data collection.
Measure: Number; unit: ratio
Arm/Group | First Open Label DCS
Number analyzed (Participants) | 1
ratio
  P50 ratio: Baseline | 44.51
  P50 ratio: Week 8 of DCS | 30

ADVERSE EVENTS:
Time Frame: 48 Weeks
Groups:
- Open Label DCS: Both participants received open label D-cycloserine (seromycin), 50 mg/d capsule, for 8 weeks.
- DCS (Crossover): Both participants received open label D-cycloserine (seromycin), 50 mg/d capsule, for 6 weeks.
- PLACEBO (CROSSOVER): Both participants received placebo for 6 weeks.
Arm/Group | Open Label DCS | DCS (Crossover) | PLACEBO (CROSSOVER) | Second Open Label DCS
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2015-04-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT02304432/ICF_000.pdf
  • Study Protocol (2015-04-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT02304432/Prot_001.pdf
  • Statistical Analysis Plan (2015-02-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT02304432/SAP_002.pdf